CLINICAL TRIAL: NCT04650347
Title: Holmium: YAG Versus Cold Knife Internal Urethrotomy in Management of Short Urethral Strictures: A Randomized Controlled Trial
Brief Title: Holmium: YAG Versus Cold Knife Internal Urethrotomy in Management of Short Urethral Strictures
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, principle investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R55/2017
Record Dates: First submitted 2020-11-24; First posted 2020-12-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Urethral Stricture, Male
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Intervention Model Description: the investigators planned to conduct a controlled trial with randomization in which eighty participants will be included with symptoms of outflow obstruction secondary to urethral stricture. this is between March 2017 and December 2019. those patients attended the outpatient clinic of our tertiary hospital of Ain Shams University. patients were allocated into 2 equal groups randomly. each group involved 40 patients. Group 1 will represent the holmium laser internal urethrotomy group while group 2 will represent the cold knife internal urethrotomy group.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: patients, data collector, and the statistician were blinded to the type of intervention. the assessment was done to group A and B
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- internal urethrotomy using Holmium laser representing group (Experimental): In group 1, a three hundred micron laser fiber was used to conduct the laser energy. holmium laser pulse energy of approximately 1 joule was used that was generated from a Holmium laser Quanta device and total power of 15 watts. the laser fiber was aimed directly to the midline at 12 o'clock position to start the procedure and cut the fibrous tissue till access to a wide lumen.
  Interventions: Procedure: visualized internal urethrotomy
- internal urethrotomy with Sachs cold knife (Active Comparator): In group B, Sache cold knife internal urethrotomy was used with the same technique as Holmium laser internal urethrotomy at the same site to mechanically cut instead of the laser fiber.
  Interventions: Procedure: visualized internal urethrotomy

INTERVENTIONS:
Procedure: visualized internal urethrotomy — incision of a urethral stricture to treat urinary obstruction using Quanta Holmium device or Sache cold knife, 18 Fr silicon catheter was kept for 7 days following the prodecure.

SUMMARY:
Urethral stricture disease is defined as narrowing of the urethral lumen because of fibrosis, which occurs in urethral mucosa and surrounding tissues. The etiology could be congenital, iatrogenic, infectious, or idiopathic.

Several techniques are currently available for minimally invasive treatment of urethral strictures, including cold-knife incision, electrocautery, and various types of laser incisions. An incision with the cold knife does not cause any thermal effect on surrounding tissues but should create a mechanical injury that may lead to recurrence in long term. An incision with the electrocautery should cause a significant thermal effect on healthy surrounding tissues resulting in recurrent strictures during follow-up. Laser treatment modalities have gained popularity in the last two decades.

the aim of this trial is to evaluate the safety and efficacy of endo-urethrotomy with Holmium laser and cold knife endo-urethrotomy

DETAILED DESCRIPTION:
Urethral stricture disease (USD) is the narrowing of the urethra from scar tissue, related to genitourinary tract infections, inflammatory skin conditions, traumatic urethral injury, pelvic radiation, and urinary tract instrumentation. It has an estimated prevalence rate of 0.6%.1-3 USD is a common and challenging problem for urologists. Multiple treatment modalities are available for the management of urethral strictures depending on the site and length of stricture, this includes simple urethral dilatation, urethral stenting, endoscopic visual internal urethrotomy (VIU), or open reconstruction.

Since 1974, Sachse's internal urethrotomy has been considered the treatment of choice for USD which is fast and simple to carry out and is associated with a short recovery time. The success rates are 33%-60%.

Bulow et al in 1979 introduced the laser for internal urethrotomy. The obvious dominance of Ho: YAG are clear vision, less bleeding, precise incision and ablation of scar tissue, and short hospital admission, however, most literature assessing the adequacy of the laser in contrast to cold-knife urethrotomy show no difference in final results.

The aim of this trial is to assess the efficacy, safety, complications, and results of Holmium laser urethrotomy and cold knife internal urethrotomy for urethral stricture.

ELIGIBILITY:
Inclusion Criteria:

* men with urethral stricture above the age of eighteen were included in our trial. the length of the urethral stricture was less than 1.5 cm.

Exclusion Criteria:

* patient with complete urethral stricture with a suprapubic catheter in place.
* patients whom internal urethrotomy is not applicable like multiple urethral strictures or balanitis xerotica obliterans.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — surgical intervention of male urethra stricture
Enrollment: 80 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum flow rate (ml/sec.) | at 3 months
  maximum flow rate, uroflow finding (ml/sec.)
Maximum flow rate(ml/sec.) | at 12 months
  maximum flow rate, uroflow finding (ml/sec.)

SECONDARY OUTCOMES:
operation time in minutes | intraoperative finding
  time of operation from cystoscopy till catheter insertion
number of patients with bleeding per urethra | first day postoperative
  postoperative bleeding around the catheter
number of patients with penile extravasation | first day postoperative
  penile swelling from fluid extravasation
number of patients with urinary tract infection | first month postoperative
  urinary tract infection from urine analysis and culture
number of patients with urethral stricture recurrence | from catheter removal up to 1 year postoperative
  recurrence of symptoms with urine outflow obstruction and difficult voiding as measured by uroflow

CONTACTS AND LOCATIONS:
Locations (1):
- Urology department - ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided